CLINICAL TRIAL: NCT05073653
Title: A Study of 68Ga-GRP PET/CT for Imaging in Low and Intermediate Risk Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202110113
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-09

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; 68Ga-GRP PET/CT; 68Ga-PSMA PET/CT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 68Ga-PSMA PET/CT Imaging (Other): Injection of the radioligand 68Ga-PSMA; Device: PET/CT; Following injection of 68Ga-PSMA, the participants will be subjected to whole body PET/CT.
  Interventions: Diagnostic Test: 68Ga-PSMA PET/CT
- 68Ga-GRP PET/CT Imaging (Other): Injection of the radioligand 68Ga-GRP; Device: PET/CT; Following injection of 68Ga-GRP, the participants will be subjected to whole body PET/CT.
  Interventions: Diagnostic Test: 68Ga-GRP PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-PSMA PET/CT — Exploratory, Single-institution Study, Comparing 68Ga-GRP PET/CT Versus 68Ga-PSMA PET/CT in Patients Diagnosed With Prostate Cancer of Low and Intermediate Risk for Radical Prostatectomy
  Arms: 68Ga-PSMA PET/CT Imaging
Diagnostic Test: 68Ga-GRP PET/CT — Exploratory, Single-institution Study, Comparing 68Ga-GRP PET/CT Versus 68Ga-PSMA PET/CT in Patients Diagnosed With Prostate Cancer of Low and Intermediate Risk for Radical Prostatectomy
  Arms: 68Ga-GRP PET/CT Imaging

SUMMARY:
Patients with primary low and intermediate risk prostate cancer (PCa) for whom radical prostatectomy are indicated, will be invited to participate to the present study.

The aim of this study is to investigate the clinical value of 68Ga-GRP positron emission tomography / computed tomography (PET/CT) compared to 68Ga-PSMA PET/CT in patients with low and intermediate risk PCa.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the second-most common cancer among men across the world, and a significant cause of death in many regions. Different stages of PCa directly affect both the therapeutic schedule and patient prognosis.

Recommended imaging modalities for initial staging include computerized tomography (CT) scan, bone scan, and Magnetic Resonance Imaging (MRI). In addition to initial work-up, Gallium-68 prostate-specific membrane antigen positron emission tomography/computer tomography (68Ga-PSMA PET/CT) is a relatively new nuclear imaging modality, showing high sensitivity and specificity. Recently, several studies have investigated the role of 68Ga-PSMA PET/CT in a first-line diagnostic setting, especially in patients with high-risk and biochemically recurrent PCa.

Therefore, PET imaging with 68Ga-PSMA may participate to optimize work-up in the staging of high-risk patients.

Another family of radiopharmaceuticals aimed to target the Gastrin-Releasing Peptide Receptor (GRP-R) which is overexpressed in early stage PCa. Various radiolabeled GRP analogues have been developed and shown encouraging results as related to the detection of primary PCa in preclinical study. However, 68Ga-GRP failed to detect some bone metastases in hormone-refractory patients. A prospective study identified that GRPR expression is not associated with Gleason score (GS) and PSMA expression, suggesting that 68Ga-GRP and 68Ga-PSMA PET/CT may be complementary in various risks of PCa diagnosis.

The aim of this pilot study is to compare 68Ga-PSMA PET/CT to 68Ga-GRP PET/CT in patients with PCa of low and intermediate risk to better understand how 68Ga-PSMA and 68Ga-GRP PET/CT could performed a primary lesion mapping and how 68Ga-PSMA and 68Ga-GRP PET/CT could be used (or combined) in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* patients divided in :

  * Patients with low risk prostate cancer (Gleason score ≤ 6 and cT1-T2a and Prostate Specific Antigen (PSA) value < 10 ng/mL);
  * Patients with intermediate risk prostate cancer (Gleason score 7 or cT2b or PSA value 10-20 ng/mL);
  * Patients with high risk prostate cancer (Gleason > 7 or cT2c or PSA value > 20 ng/mL);
  * Candidate for radical prostatectomy after discussion in multidisciplinary committee;
  * Written informed consent willingly obtained.

Exclusion Criteria:

* Any kind of previous treatment for prostate cancer (hormonal treatment, EBRT, brachytherapy, cryotherapy, etc…);
* Patient not candidate for radical prostatectomy and/or unable to benefit from surgery;
* Patient under legal protection or unable to express its own consent;
* Patient within exclusion period from another clinical trial;
* Claustrophobia (unable to accept PET/CT scanning).

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-10-11 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Median Standardized Uptake Value (SUV) | Day 0 (inclusion) or Day 2 to 21
  Median Standardized Uptake Value (SUV) of 68Ga-GRP
Median Standardized Uptake Value (SUV) | Day 0 (inclusion) or Day 2 to 21
  Median Standardized Uptake Value (SUV) of 68Ga-PSMA

SECONDARY OUTCOMES:
Gleason score of lesion reported from pathological findings | Day 3 to 60
  Gleason score was used to rank prostate cancer risk and was associated with SUV
Immunoreactive of lesion | Day 3 to 60
  Immunoreactive analysis of PSMA and GRPR

OTHER OUTCOMES:
Correlation analysis between SUV and Gleason score | Day 3 to 60
  Correlation analysis

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Hu, PhD, MD, Study Director — Department of PET Center,Xiangya Hospital,Central South University
Locations (1):
- Department of PET Center,Xiangya Hospital,Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Result] Fenton JJ, Weyrich MS, Durbin S, Liu Y, Bang H, Melnikow J. Prostate-Specific Antigen-Based Screening for Prostate Cancer: Evidence Report and Systematic Review for the US Preventive Services Task Force. JAMA. 2018 May 8;319(18):1914-1931. doi: 10.1001/jama.2018.3712. PMID 29801018
- [Result] Perera M, Papa N, Roberts M, Williams M, Udovicich C, Vela I, Christidis D, Bolton D, Hofman MS, Lawrentschuk N, Murphy DG. Gallium-68 Prostate-specific Membrane Antigen Positron Emission Tomography in Advanced Prostate Cancer-Updated Diagnostic Utility, Sensitivity, Specificity, and Distribution of Prostate-specific Membrane Antigen-avid Lesions: A Systematic Review and Meta-analysis. Eur Urol. 2020 Apr;77(4):403-417. doi: 10.1016/j.eururo.2019.01.049. Epub 2019 Feb 14. PMID 30773328
- [Result] Mansi R, Fleischmann A, Macke HR, Reubi JC. Targeting GRPR in urological cancers--from basic research to clinical application. Nat Rev Urol. 2013 Apr;10(4):235-44. doi: 10.1038/nrurol.2013.42. Epub 2013 Mar 19. PMID 23507930
- [Result] Wieser G, Mansi R, Grosu AL, Schultze-Seemann W, Dumont-Walter RA, Meyer PT, Maecke HR, Reubi JC, Weber WA. Positron emission tomography (PET) imaging of prostate cancer with a gastrin releasing peptide receptor antagonist--from mice to men. Theranostics. 2014 Feb 1;4(4):412-9. doi: 10.7150/thno.7324. eCollection 2014. PMID 24578724
- [Result] Zhang J, Niu G, Fan X, Lang L, Hou G, Chen L, Wu H, Zhu Z, Li F, Chen X. PET Using a GRPR Antagonist 68Ga-RM26 in Healthy Volunteers and Prostate Cancer Patients. J Nucl Med. 2018 Jun;59(6):922-928. doi: 10.2967/jnumed.117.198929. Epub 2017 Nov 9. PMID 29123014
- [Result] Touijer KA, Michaud L, Alvarez HAV, Gopalan A, Kossatz S, Gonen M, Beattie B, Sandler I, Lyaschenko S, Eastham JA, Scardino PT, Hricak H, Weber WA. Prospective Study of the Radiolabeled GRPR Antagonist BAY86-7548 for Positron Emission Tomography/Computed Tomography Imaging of Newly Diagnosed Prostate Cancer. Eur Urol Oncol. 2019 Mar;2(2):166-173. doi: 10.1016/j.euo.2018.08.011. Epub 2018 Sep 22. PMID 31017093